CLINICAL TRIAL: NCT04316182
Title: A Phase II triAl of Cabozantinib for hepaTocellular carcInoma Patients intOlerant to Sorafenib Treatment or First Line Treatment Different to sorafeNib. (ACTION Trial)
Brief Title: Cabozantinib in Patients With Hepatocellular Carcinoma (ACTION)
Acronym: ACTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTION; 2019-004991-20 (EudraCT Number)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Cabozantinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib at 60 mg/day in monotherapy until symptomatic tumor progression, unacceptable adverse events, patient decision or death
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib 60 mg/day. Cabozantinib dose will be modified upon development of adverse events.
  Other Names: Cabometix

SUMMARY:
Cabozantinib, a small molecule directed to vascular endothelial growth factor receptors, MET and AXL, has shown to significantly improve the overall survival (OS) over placebo in the randomized phase 3 CELESTIAL trial in patients who had up to two lines of prior systemic therapy (including sorafenib) with progression on at least one in comparison to patients who received best supportive care.

Although cabozantinib shares similar targets with sorafenib/regorafenib, they present different toxicity profile. While the most common grade 3-4 Adverse Events reported for sorafenib were fatigue (4%), diarrhea (8%), hand-foot reaction (8%) and hypertension (2%); the most frequent grade 3-4 Adverse Events for cabozantinib were hand-foot reaction (3.6%), hypertension (3.4%) and elevation of AST (2.6%).

In clinical practice, regorafenib, ramucirumab and cabozantinib are approved by European Medicines Agency (EMA) as second-line treatment approved by EMA until now. However, more than 40% of candidate patients to 2nd line do not meet the RESORCE criteria or REACH-2 trial and are only candidates to cabozantinib treatment. However, investigators do not have safety data about those patients who are treated with other treatments than sorafenib in first line neither data about the real impact of sorafenib-intolerant patients according to the RESORCE trial definition.

For this reason, investigators propose to explore the role of cabozantinib in patients who were not considered in the CELESTIAL trial.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular Carcinoma (HCC) diagnosed according to criteria of American Association for the Study of Liver Diseases (AASLD) definition in 2010.
2. Intolerant to sorafenib according to RESORCE trial definition or patients who received treatment different to sorafenib as first-Line treatment.
3. The subject has disease that is not amenable to a curative treatment approach (eg, transplant, surgery, radiofrequency ablation)
4. Recovery to ≤ Grade 1 according to (CTCAE) v.5.0. from toxicities related to any prior treatments, unless the adverse events are clinically non-significant and/or stable on supportive therapy
5. Respect the 15 days of first-line treatment washout before starting cabozantinib
6. Age ≥ 18 years old on the day of consent
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Adequate hematologic function, based upon meeting the following laboratory criteria within 7 days before starting therapy:

   1. absolute neutrophil count (ANC) ≥ 1200/mm3 (≥ 1.2 x 10*9/L)
   2. platelets ≥ 60,000/mm3 (≥ 60 x 10*9/L)
   3. hemoglobin ≥ 8 g/dL (≥ 80 g/L)
9. Adequate renal function, based upon meeting the following laboratory criteria within 7 days before starting therapy:

   1. Serum creatinine ≤ 1.5 × upper limit of normal or calculated creatinine clearance ≥ 40 mL/min (using the Cockcroft-Gault equation) AND
   2. Urine protein/creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol) or 24-hour urine protein < 1 g
10. Child-Pugh Score of A
11. Total bilirubin ≤ 2 mg/dL (≤ 34.2 μmol/L) within 7 days before starting therapy
12. Serum albumin ≥ 2.8 g/dL (≥28 g/L) within 7 days before starting therapy
13. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5.0 upper limit of normal (ULN) within 7 days before starting therapy
14. Hemoglobin A1c (HbA1c) ≤ 8% within 28 days before starting therapy (if HbA1c results are unavailable [eg, hemoglobin variant], a fasting serum glucose ≤ 160 mg/dL)
15. Antiviral therapy per local standard of care if active hepatitis B (HBV) infection
16. Capable of understanding and complying with the protocol requirements and signed informed consent
17. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment
18. Female subjects of childbearing potential must not be pregnant at screening.
19. Subjects must consent to perform a tumor liver biopsy within 4 weeks before starting cabozantinib, allowing the acquisition of a tumor sample for performance of correlative studies.

Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
2. Radiation therapy (eg, I-131 or Y-90) within 4 weeks (2 weeks for radiation for bone metastases or radionuclide treatment within 6 weeks of starting therapy) (subject is excluded if there are any clinically relevant ongoing complications from prior radiation therapy)
3. Prior cabozantinib treatment
4. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before starting therapy. Eligible subjects must be without corticosteroid treatment at the time of starting therapy.
5. Concomitant anticoagulation, at therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, low molecular weight heparin (LMWH), thrombin or coagulation factor X (FXa) inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin for cardioprotection (per local applicable guidelines), low-dose warfarin (≤ 1 mg/day), and low dose LMWH are permitted.
6. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions

   a. Cardiovascular disorders including:

   i. Symptomatic congestive heart failure, unstable angina pectoris, or serious cardiac arrhythmias ii. Uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic, or 100 mm Hg diastolic despite optimal antihypertensive treatment iii. Stroke (including TIA), myocardial infarction, or another ischemic event within 6 months before starting therapy iv. Thromboembolic event within 3 months before starting therapy. Subjects with thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor are eligible

   b. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

   i. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before starting therapy iii. Note: Complete healing of an intra-abdominal abscess must be confirmed prior to starting therapy

   c. Major surgery within 2 months before starting therapy. Complete healing from major surgery must have occurred 1 month before starting therapy. Complete healing from minor surgery (eg, simple excision, tooth extraction) must have occurred at least 7 days before starting therapy. Subjects with clinically relevant complications from prior surgery are not eligible

   d. Cavitating pulmonary lesion(s) or endobronchial disease

   e. Lesion invading a major blood vessel including, but not limited to: pulmonary artery, or aorta. Subjects with lesions invading the portal vasculature are eligible.

   f. Clinically significant bleeding risk including the following within 3 months of starting therapy: hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors

   g. Other clinically significant disorders such as:

   i. Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS)-related illness. Subjects with active hepatitis virus infection controlled with antiviral therapy are eligible.

   ii. Serious non-healing wound/ulcer/bone fracture iii. Malabsorption syndrome iv. Uncompensated/symptomatic hypothyroidism v. Requirement for hemodialysis or peritoneal dialysis vi. History of solid organ transplantation
7. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding. Subjects treated with adequate endoscopic therapy (according to institutional standards) without any episodes of recurrent GI bleeding requiring transfusion or hospitalization for at least 6 months prior to study entry are eligible.
8. Moderate or severe ascites. Note that controlled ascites with stable dose of diuretics in the last month is allowed.
9. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 7 days before starting therapy
10. Inability to swallow tablets
11. Previously identified allergy or hypersensitivity to components of the study treatment formulations
12. Pregnant or lactating females
13. Diagnosis of another malignancy within 2 years before starting therapy, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy
14. History of allergy to study drug components.
15. Prisoners or subjects who are involuntarily incarcerated
16. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg. infectious disease) illness
17. Inability to comply with restrictions and prohibited activities/treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Reig, MD, Principal Investigator — BCLC group. Liver Unit. Hospital Clinic. Ciberehd
Locations (6):
- Spain (6):
  - Hospital Clinic, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Institut Català D'Oncologia - Hospital Duran I Reynals, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Central de Asturias, Oviedo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.67 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  Latin or Hispanic | 1
  White | 22
Tumor burden [Count of Participants; unit: Participants]
  Extrahepatic spread | 3
  Multinodular | 14
  Portal invasion | 4
  Single or up to 3 nodules >= 3cm | 3
Cirrhosis [Count of Participants; unit: Participants] | 19
Vascular Invasion [Count of Participants; unit: Participants] | 8
ECOG [Count of Participants; unit: Participants]
  ECOG 0: Fully active, able to carry on all pre-disease performance without restriction | 20
  ECOG 1: Restricted in strenuous activity but ambulatory/able to carry out work of light nature | 4
First line treatment [Count of Participants; unit: Participants]
  Atezolizumab+bevacizumab | 3
  Lenvatinib | 1
  Nivolumab+ipilimumab | 1
  Sorafenib | 18
  Tislelizumab | 1
Worst type of progression [Count of Participants; unit: Participants]
  Extrahepatic growth | 2
  Intrahepatic growth | 8
  New extrahepatic lesion | 1
  New intrahepatic lesion | 11
  Not available | 2
Worst first progression pattrern [Count of Participants; unit: Participants]
  Extrahepatic growth | 2
  Intrahepatic growth | 7
  New extrahepatic lesion | 3
  New intrahepatic lesion | 10
  Not available | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adverse Events (AE) ≥ Grade 3 (CTCAE 5.0) Excluding Palmar-plantar Erythrodysesthesia
Description: Percentage of patients with Grade 3 AEs in relation with total number of treated patients
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Participants | 16

2. Primary Outcome: Rate of Adverse Events
Description: Percentage of patients with AEs in relation with total number of treated patients
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Participants | 24

3. Primary Outcome: Rate of Related-AEs
Description: Percentage of patients with related AEs in relation with total number of treated patients
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Participants | 24

4. Primary Outcome: Rate of Death Due to Adverse Events
Description: Percentage of patients who die during treatment due to adverse events in relation with total number of treated patients
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Participants | 0

5. Primary Outcome: Rate of AEs Leading to Treatment Discontinuation
Description: Percentage of patients with AEs leading to treatment discontinuation in relation with total number of treated patients
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
Participants | 3

6. Secondary Outcome: Time to Progression (TTP)
Description: Time from the date of start of treatment until the date of objective disease progression or death
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
months | 6 [3 to 8]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the number of subjects with a best overall response of a complete response (CR) or partial response (PR) divided by the number of included patients
Time Frame: Up to 18 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
percentage of patients | 8.3 [1.0 to 27.0]

8. Secondary Outcome: Pattern of Progression
Description: Type of progression divided by number of patients
Time Frame: Up to 18 months
Population: They are included patients with available radiological progression (18 patients). One patient did not progress and 5 patients died due to progression without having a corresponding radiological evaluation.
Measure: Number; unit: percentage of patients
Arm/Group | Cabozantinib
Number analyzed (Participants) | 18
percentage of patients
  Intrahepatic growth (IHG) | 44.4
  New intrahepatic lesion (NIH) | 22.2
  Extrahepatic growth (EHG) | 11.1
  New extrahepatic lesion (NEH) | 22.2

9. Secondary Outcome: Overall Survival (OS)
Description: Time from the date of start of treatment until the date of death
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
months | 11 [8 to 20]

10. Secondary Outcome: Post-progression Survival (PPS)
Description: Time from the date of disease progression until the date of death
Time Frame: Up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
months | 5 [2 to NA] — The statistical program does not provide the upper limit of the interval for this outcome due to insufficient number of participants with the event.

11. Secondary Outcome: Rate of Patients Who Develop New Extra-hepatic Spread
Description: Number of subjects who develop new extra-hepatic spread divided by number of included patients
Time Frame: Up to 18 months
Measure: Number; unit: percentage of patients
Arm/Group | Cabozantinib
Number analyzed (Participants) | 24
percentage of patients | 22

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated at each study visit through treatment completion and 30 days after the last dose, an average of 34 weeks.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 15/24
Serious Adverse Events (participants affected / at risk) | 8/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=24)
Pyrexia (General disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=24)
Hypertension (Vascular disorders) | 16 (27)
Asthenia (General disorders) | 6 (21)
Discomfort (General disorders) | 2 (2)
Fatigue (General disorders) | 12 (17)
Mucosal inflammation (General disorders) | 3 (3)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 2 (2)
Decreased appetite (General disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (16)
Aspartate aminotransferase increased (Investigations) | 6 (13)
Blood bilirubin increased (Investigations) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (5)
Joint injury (Injury, poisoning and procedural complications) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Tension headache (Nervous system disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Ascites (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 12 (31)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 5 (6)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 3 (5)
Jaundice (Hepatobiliary disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 15 (46)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT04316182/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT04316182/SAP_001.pdf